CLINICAL TRIAL: NCT01006070
Title: Prospective Observation Study of Health-related QOL, Physical Function & Respiratory Function in Patients w/ Myeloma Affecting Spine: The Impact of Disease,Fractures & Effect of Vertebral Augmentation w/ Kyphoplasty
Brief Title: Health-Related Quality of Life (QOL), Physical and Respiratory Function in Patients With Myeloma Affecting the Spine
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Medtronics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0901Wolf
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; spinal disease
MeSH Terms: conditions — Multiple Myeloma; Spinal Diseases | interventions — Kyphoplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with existing spinal fractures: Myeloma patients with documented x-ray evidence of spinal fractures.
  Interventions: Procedure: kyphoplasty
- Patients without spinal fractures: Myeloma patients with bony disease in the spine without existing fractures.
  Interventions: Procedure: kyphoplasty

INTERVENTIONS:
Procedure: kyphoplasty — surgical kyphoplasty
  Other Names: balloon kyphoplasty

SUMMARY:
The purpose of this study is to create a prospective database of patients with myeloma affecting the spine. This database will define changes in health-related quality of life over time, and the effect of incident fractures and their treatment on specific measures of pain, physical function, pulmonary function, and future fractures. In 2008, the UCSF Myeloma Service was actively caring for 347 patients with myeloma, of which 150 patients had lytic lesions on radiographs, and 100 had a known vertebral fracture. This population, as well as any new myeloma patients, will serve as the source of the study population.

DETAILED DESCRIPTION:
The UCSF Adult Hematology Program maintains a data base of all patients with a diagnosis of multiple myeloma seen in the Clinic. As patients are treated, relapse, receive new treatment, are transplanted, or pass away, these data are entered into this Multiple Myeloma Data Base (MMDB).

The MMDB will be expanded to include parameters to identify those patients with myeloma affecting the spine. A recruitment letter will be sent to all patients in the MMDB identified as having myeloma affecting the spine asking if they would be interested in participating in this study.

Patients who agree to participate in the study will be given an appointment to meet with Dr. Wolf or Dr. Martin to discuss the study and if willing, to sign the informed consent document. They will have an exam and history taken that includes fracture history.

Patients who have signed consent will be sent for thoracic-lumbar spine films (unless they had prior spine films taken within the last 3 months). Those with normal films will not be eligible to be enrolled to the study. Those with abnormal spinal films will then be sent for MRI of the spine, pulmonary function testing, and meeting with Dr. R. Yonge who will administer the various QOL tests described below.

All eligible established and new patients will be invited to participate in the prospective study. Patients who sign the informed consent will be included in the prospective study. A minimum of 25 patients with vertebral fractures and 25 patients without fractures, will be observed to measure the impact of fractures on health-related quality of life. Study enrollment will be complete when 25 patients without a new fracture and 25 patients with a new fracture treated by balloon kyphoplasty have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of Multiple Myeloma and evidence of myelomatous lesions in the spine, including plasmacytomas, lytic lesions and fractures.

Exclusion Criteria:

* Myeloma patients without evidence of bony lesions in the spine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multiple myeloma patients with spinal lesions
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Identify and prospectively study patients with myeloma affecting the spine, with or without compression fractures. Use standardized tools to assess health-related QOL, physical and respiratory function in these patients | 1 year

SECONDARY OUTCOMES:
Measure: effect of pre-existing spinal fracture, prospectively measure effect of fractures and treatment on QOL, physical and respiratory function, and incidence of future fractures | 1 year
Identify x-ray predictors of future/pending vertebral fractures | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wolf, MD, Principal Investigator — University of California, San Francisco; Sigurd Berven, MD, Principal Investigator — University of California, San Francisco; Thomas Martin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States